CLINICAL TRIAL: NCT00957905
Title: A Non-randomized Phase 2 Study of Alvocidib (Flavopiridol) Plus Oxaliplatin With or Without 5-FU and Leucovorin for Relapsed or Refractory Germ-Cell Tumors
Brief Title: Alvocidib and Oxaliplatin With or Without Fluorouracil and Leucovorin Calcium in Treating Patients With Relapsed or Refractory Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01405; NCI-2011-01405 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSKCC-09034; CDR0000646950; 09-034 (Other: Memorial Sloan-Kettering Cancer Center); 8258 (Other: CTEP); N01CM00071 (NIH); N01CM62206 (NIH); P30CA008748 (NIH); U01CA062491 (NIH); U01CA062505 (NIH); U01CA069856 (NIH); U01CA069912 (NIH); U01CA099168 (NIH)
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Recurrent Extragonadal Seminoma; Recurrent Malignant Extragonadal Germ Cell Tumor; Recurrent Malignant Extragonadal Non-Seminomatous Germ Cell Tumor; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Ovarian Germ Cell Tumor; Stage III Testicular Cancer; Stage IV Extragonadal Non-Seminomatous Germ Cell Tumor; Stage IV Extragonadal Seminoma; Stage IV Ovarian Germ Cell Tumor
MeSH Terms: conditions — Testicular Neoplasms | interventions — cytokine inducible SH2-containing protein; alvocidib; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin

ARMS (2):
- Part A (alvocidib and oxaliplatin) (Experimental): Patients receive alvocidib IV over 1 hour and oxaliplatin IV over 2 hours on days 1, 15, and 29. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alvocidib Hydrochloride; Drug: Oxaliplatin
- Part B (alvocidib and FOLFOX) (Experimental): Patients receive alvocidib IV over 1 hour, oxaliplatin IV over 2 hours, and leucovorin calcium IV over 2 hours followed by fluorouracil IV continuously over 48 hours on days 1, 15, and 29. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alvocidib Hydrochloride; Drug: Fluorouracil; Drug: Leucovorin Calcium; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Alvocidib Hydrochloride — Given IV
  Other Names: 4H-1-Benzopyran-4-one, 2-(2-chlorophenyl)-5, 7-dihydroxy-8-(3-hydroxy-1-methyl-4-piperidinyl)-, hydrochloride, (-)-cis-; Flavopiridol Hydrochloride; HL-275; HMR 1275; L-86-8275; L-868275; MDL 107,826A; MDL-107826A
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Actino-Hermal; Adrucil; Arumel; Cytosafe; Efudex; Efurix; Fiverocil; Fluoro Uracil; Fluoroplex; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Flurox; Ribofluor; Ro 2-9757; Ro-2-9757; Timazin
  Arms: Part B (alvocidib and FOLFOX)
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Part B (alvocidib and FOLFOX)
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669

SUMMARY:
This phase II trial is studying alvocidib and oxaliplatin to see how well they work when given with or without fluorouracil and leucovorin calcium in treating patients with relapsed or refractory germ cell tumors. Drugs used in chemotherapy, such as alvocidib, oxaliplatin, fluorouracil, and leucovorin calcium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving alvocidib together with oxaliplatin with or without fluorouracil and leucovorin calcium may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the antitumor efficacy of the combination of flavopiridol and oxaliplatin with or without 5-FU and leucovorin in patients with relapsed or refractory GCT. The necessity of 5-FU and leucovorin to the combination will also be indirectly tested in this study.

SECONDARY OBJECTIVES:

I. To further evaluate the safety of flavopiridol in combination with oxaliplatin with or without 5-fluorouracil and leucovorin in patients with refractory or relapsed GCT.

II. To evaluate the time to tumor response (TTR) and progression-free survival for patients with refractory or relapsed GCT treated with flavopiridol in combination with oxaliplatin with or without 5-fluorouracil and leucovorin.

III. To explore the association between treatment response and p21, p53 and apoptotic markers.

OUTLINE: Patients are initially enrolled in part A (closed to accrual as of 11/15/2010). Depending on response to treatment, additional patients may be enrolled in part B.

PART A (alvocidib and oxaliplatin) (closed to accrual as of 11/15/2010): Patients receive alvocidib IV over 1 hour and oxaliplatin IV over 2 hours on days 1, 15, and 29. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

PART B (alvocidib and FOLFOX): Patients receive alvocidib IV over 1 hour, oxaliplatin IV over 2 hours, and leucovorin calcium IV over 2 hours followed by fluorouracil IV continuously over 48 hours on days 1, 15, and 29. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity. Tumor tissue samples may be collected periodically for further laboratory analysis.

After completion of study treatment, patients are followed up every 4-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed germ cell tumor (GCT)

  * Seminoma or non-seminoma
* Progressive disease after prior cisplatin-based therapy AND meets 1 of the following criteria:

  * Not considered to be a candidate for potentially curative therapy
  * Previously treated with high-dose chemotherapy regimens
  * Does not wish to undergo potentially curative high-dose therapy
* Measurable or evaluable disease, as defined by 1 of the following criteria:

  * Unidimensionally measurable metastatic disease, defined as ≥ 1 malignant tumor mass that can be accurately measured in ≥ 1 dimension as ≥ 20 mm by conventional CT scan or MRI or as ≥ 10 mm by spiral CT scan

    * Bone lesions, ascites, peritoneal carcinomatosis, miliary lesions, pleural or pericardial effusions, lymphangitis of the skin or lung, cystic lesions, or irradiated lesions are not considered measurable disease
    * Patients with measurable disease only (i.e., normal tumor markers) must have ≥ 1 site of disease that has not been previously irradiated
  * Elevation of alpha-fetoprotein > 15 ng/mL and/or elevation of beta-human chorionic gonadotropin > 2.2 mIU/L

    * If tumor markers are not elevated, ≥ 1 site of measurable disease must be present
* No known untreated CNS metastasis or primary CNS tumor

  * Patients who have undergone local treatment for brain metastases and whose brain metastases are demonstrated to be stable by repeat imaging studies performed ≥ 4 weeks after treatment are eligible
* Karnofsky performance status 70-100%
* ANC ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Serum creatinine ≤ 2.0 times upper limit of normal (ULN)
* Total serum bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN (unless elevation is due to underlying malignancy)
* Not pregnant or nursing
* Negative pregnancy test by ultrasound
* Fertile patients must use effective contraception
* Willing and able to comply with scheduled study visits, treatment plans, laboratory tests, follow-up tests for safety or effectiveness, and other study procedures
* Mediport or Broviac access required for patients enrolled in part B of the study
* No serious active infections
* No significant (≥ grade 2) or persistent ongoing toxicity, including peripheral neuropathy, from prior therapy
* None of the following within the past 6 months:

  * Myocardial infarction
  * Severe/unstable angina
  * Coronary/peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
* No contraindication to any of the study drugs
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, interfere with the interpretation of study results, and, in the judgement of the investigator, may make the patient inappropriate for study entry
* No concurrent anti-retroviral therapy for HIV-positive patients
* Recovered from prior radiotherapy or surgery

  * Residual grade 1 toxicities allowed
* No prior alvocidib
* At least 2 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C), immunotherapy, or radiotherapy
* More than 4 weeks since prior major surgery
* No other concurrent approved or investigational anticancer treatment, including surgery, radiotherapy, chemotherapy, biologic-response modifiers, hormone therapy, or immunotherapy
* No concurrent participation in another investigational treatment clinical trial

  * Concurrent participation in supportive care trials or non-treatment trials (e.g., quality of life or laboratory analysis studies) allowed
* No concurrent vitamins, antioxidants, herbal preparations, or supplements, except for a single-tablet multivitamin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Riverview Hospital, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: 6 weeks: Flavopiridol: 70 mg/m2/day IV over 1 hr on days 1, 15 and 29. Oxaliplatin: 85 mg/m2/day IV over 2 hrs on days 1, 15 and 29.
- Part B: 6 wks: Flavopiridol:70 mg/m2/day IV 1 hr Days 1, 15 & 29. Oxaliplatin:85 mg/m2/day IV 2 hrs Days 1, 15 & 29. Leucovorin:400 mg/m2/day IV 2 hrs Days 1, 15 & 29.
  5-FU: 400 mg/m2 IV 15 min, and 1800 mg/m2 IV 48 hrs Days 1-2, 15-16 & 29-30.
Period: Part A
Arm/Group | Part A | Part B
Started | 7 | 0
Completed | 7 | 0
Not Completed | 0 | 0
Period: Part B
Arm/Group | Part A | Part B
Started | 0 | 29
Completed | 0 | 25
Not Completed | 0 | 4
Not completed — Not Treated | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A (Alvocidib and Oxaliplatin) | Part B (Alvocidib and FOLFOX) | Total
Number analyzed (Participants) | 7 | 29 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 29 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 7 | 28 | 35
Region of Enrollment [Number; unit: participants]
  United States | 7 | 29 | 36

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Number of Participants with Partial Response (PR), Stable Disease (SD), Progression of Disease (POD) Per Response Evaluation Criteria In Solid Tumors Criteria" (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (POD); POD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Within 3 courses of treatment
Measure: Number; unit: participants
Arm/Group | Part A (Alvocidib and Oxaliplatin) | Part B (Alvocidib and FOLFOX)
Number analyzed (Participants) | 7 | 25
participants
  Partial Response | 0 | 6
  Stable Disease | 2 | 10
  Progression of Disease | 5 | 9

2. Other Pre Specified Outcome: Toxicity
Description: graded using the NCI CTCAE version 4.0.See adverse event section
Time Frame: Up to 4 years
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Progression-free Survival
Time Frame: From treatment start until first documented progression or death, assessed up to 4 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Time to Tumor Response
Time Frame: From treatment start until first documented CR or PR, assessed up to 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Part A (Alvocidib and Oxaliplatin) | Part B (Alvocidib and FOLFOX)
Serious Adverse Events (participants affected / at risk) | 4/7 | 7/29
Other Adverse Events (participants affected / at risk) | 5/7 | 23/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (Alvocidib and Oxaliplatin) (N=7) | Part B (Alvocidib and FOLFOX) (N=29)
Fever (General disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decrease (Investigations) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (Alvocidib and Oxaliplatin) (N=7) | Part B (Alvocidib and FOLFOX) (N=29)
Alkaline phosphatase increased (Investigations) | 2 (5) | 2 (7)
Anemia (Blood and lymphatic system disorders) | 2 (18) | 8 (46)
Blood bilirubin increased (Investigations) | 1 (3) | 0 (0)
Creatinine increased (Investigations) | 1 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 5 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 4 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (12) | 6 (16)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (13) | 6 (15)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (10) | 10 (39)
Neutrophil count decreased (Investigations) | 1 (1) | 12 (39)
Platelet count decreased (Investigations) | 2 (3) | 17 (60)
White blood cell decreased (Investigations) | 2 (6) | 12 (55)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 4 (6)
INR increased (Investigations) | 0 (0) | 2 (7)
Nausea (Gastrointestinal disorders) | 0 (0) | 8 (12)
Vomiting (Gastrointestinal disorders) | 0 (0) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less